CLINICAL TRIAL: NCT00551499
Title: Cardiac Resynchronisation Therapy in Combination With Overdrive Pacing in the Treatment of Central Sleep Apnea in CHF
Acronym: Morpheus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 113
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Central Sleep Apnea
Keywords: Sleep Apnea, CRT
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Central; Sleep Apnea Syndromes; Creatine deficiency, X-linked

STUDY DESIGN:
Intervention Model Description: Comparing effect of CRT in patients with and without CSA + comparing effect of AOP in combination with CRT in patients with CSA
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRT for patients with CSA (No Intervention): Patients suffering from HF with central Sleep Apnea (CSA) programmed to DDD/45 (CRT) for 12 weeks. Intervention is CRT.
- CRT + AOP for patients with CSA (Active Comparator): Patients suffering from HF with central Sleep Apnea programmed to DDD/+15 bpm nocturnal rate (CRT + AOP) for 12 weeks. Intervention is the AOP in addition to CRT.
  Interventions: Device: CRT + AOP

INTERVENTIONS:
Device: CRT + AOP — The CSA group will undergo 2 sleep evaluation on two consecutive nights, during which the device will be programmed according to the randomization scheme (one night CRT, DDD/45 and the other CRT, DDD/15 bpm over mean nocturnal heart rate). The mean nocturnal heart rate over the last week is derived from the device memory.
  Arms: CRT + AOP for patients with CSA

SUMMARY:
The primary objective of this study is to compare the Apnea- Hypopnea Index in HF patients with concomitant CSA, after 12 weeks of CRT alone to CRT in combination with one night of overdrive pacing. Secondary objectives are to evaluate the effects of a single night of overdrive pacing applied after 12 weeks of CRT vs. CRT alone on breathing events, sleeping events, and neurohormonal markers. An additional secondary objective of the study is to compare the efficacy of CRT in HF patients with concomitant CSA to HF patients without concomitant CSA.

DETAILED DESCRIPTION:
Sleep apnea is a common and often undiagnosed disorder associated with substantial cardiovascular morbidity and mortality. In recent years studies have been published presenting the relationship between heart failure (HF) and central sleep apnea (CSA). CSA associated with Cheyne-Stokes respiration is a form of periodic breathing in which central apneas and hypopnea alternate with periods of hyperventilation, characterized by a regular crescendo-decrescendo oscillation of tidal volume, which is thought to be caused by dysfunction of central respiratory control. Unlike, obstructive sleep apnea (OSA), CSA likely arises as a consequence of HF.Since 2002, several results have reported on the benefit of atrial overdrive (AOP) pacing in patients suffering from sleep apnea. These results could not be confirmed for obstructive sleep apnea in several subsequent studies. Cardiac resynchronization therapy (CRT) has been proposed as another potential therapeutic pacing approach for CSA by two recently published investigations.The combined therapeutic impact of AOP and CRT (CRT+AOP) so far has not been investigated.We aimed to evaluate the effect of CRT alone and CRT+AOP on CSA in patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented clinical history of symptomatic but stable congestive heart failure, NYHA III or NYHA IV, of at least six weeks duration.
* Patient has an indication for a CRT device, or patients with previous pacemaker indication, except Sick Sinus Syndrome, and currently in need for an upgrade to a CRT device
* Patient is scheduled for the implantation of a CRT device
* Patient is over 18 years of age
* Patient provides Informed Consent

Exclusion Criteria:

* Inability to complete overnight sleep study as specified by the protocol
* Myocardial infarction or coronary revascularization procedure within 2 calendar months prior to enrollment
* Planned or strong likelihood of cardiac surgery within 4 months following enrollment
* A spirometric confirmation of obstructive lung disease
* Evidence of obstructive sleep apnea at baseline polysomnography
* Body mass index >30 kg/m²
* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
AHI | 12 weeks
  To demonstrate that a single night of overdrive pacing applied after 12 weeks of cardiac resynchronization therapy in comparison to cardiac resynchronization alone will improve sleep apnea as measured by Apnea- hypopnea- index (AHI)

SECONDARY OUTCOMES:
NYHA class | 12 weeks
  To evaluate the effects of nocturnal overdrive pacing applied after 12 weeks of CRT vs. CRT alone on NYHA
Echocardiographic parameter | 12 weeks
  To evaluate the effects of nocturnal overdrive pacing applied after 12 weeks of CRT vs. CRT alone on LVEF
Neurohormonal parameter | 12 weeks
  To evaluate the effects of nocturnal overdrive pacing applied after 12 weeks of CRT vs. CRT alone on neurohormonal marker NT pro-BNP
Clinical parameter | 12 weeks
  To evaluate the effects of nocturnal overdrive pacing applied after 12 weeks of CRT vs. CRT alone on the clinical parameter VO2max
Quality of Life | 12 weeks
  To evaluate the effects of nocturnal overdrive pacing applied after 12 weeks of CRT vs. CRT alone on Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: S Andreas, Prof. Dr, Principal Investigator — Georg-August-Universität, Göttingen, Department of Cardiology and Pneumology, Robert-Koch Str. 40, 37075 Göttingen, Germany
Locations (2):
- Germany (2):
  - Medizinische Klinik und Poliklinik II Universitätsklinikum, University of Bonn, Bonn
  - Georg-August-Universität, Department of Cardiology and Pneumology, Göttingen